CLINICAL TRIAL: NCT07117760
Title: Prospective Clinical Trial of Low-dose 225Ac-LNC1011 in the Treatment of Metastatic Castration-Resistant Prostate Cancer
Brief Title: Prospective Clinical Trial of 225Ac-LNC1011 in the Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstAHFujian-225Ac-LNC1011
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 225Ac-LNC1011 (Experimental): Participant will receive 3.7 MBq (+/- 10%) 225Ac-LNC1011, once every 8-10 weeks for a planned 4 cycles
  Interventions: Drug: 225Ac-LNC1011; Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 225Ac-LNC1011 — administered intravenously once every 8-10 weeks (1 cycle) for 4 cycles
Drug: 68Ga-PSMA-11 — Intravenous dose of approx. 150 MBq at screening and at time of centrally confirmed radiographic progressive disease

SUMMARY:
PSMA is an ideal target for precision diagnosis and treatment of prostate cancer. LNC1011 is a novel albumin-binding PSMA-targeted radioligand. This study aims to explore the safety and efficacy of 225Ac-labeled LNC1011 for treating patients with PSMA-positive metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA)-targeted radioligand therapy has demonstrated promising potential in treating metastatic castration-resistant prostate cancer (mCRPC). Modification of PSMA radioligans with albumin-binding motifs prolonging blood circulation significantly enhances tumor uptake and therapeutic efficacy. LNC1011 incorporates dansylated amino acids as a novel, relatively weaker and superior albumin binder, achieving a refined balance between increased tumor accumulation, safety, and diagnostic performance. This enables a unified theranostic approach within a single molecular framework.

Alpha-emitting radionuclide therapeutics offer unique advantages for cancer treatment. Regarding tumoricidal effects: Alpha emitters generate alpha particles during decay, possessing a linear energy transfer (LET) nearly 100 times higher than beta emitters, resulting in significantly superior tumor eradication. Beta emitters primarily cause single-strand DNA breaks, potentially allowing tumor cell repair and recurrence. In contrast, alpha emitters directly induce irreparable double-strand DNA breaks, leading to permanent tumor cell kill. This has earned them the designation "surgical knife-like radiotherapy." Furthermore, clinical trial data indicate that alpha emitters can trigger tumor immune responses while killing cancer cells, demonstrating synergistic effects with immunotherapy and achieving a "1 + 1 > 2" outcome in cancer therapy. Regarding safety: Alpha particles have an extremely short range (a few cell diameters), causing minimal damage to surrounding normal tissues with almost negligible side effects, thus offering superior safety. Actinium-225 has a half-life of 9.92 days. During this period, it decays through a series of alpha and beta decays, maximizing its therapeutic potential.

In this single-arm study, we will investigate the safety and efficacy of low-dose 225Ac-LNC1011 for the treatment of mCRPC. 225Ac-LNC1011 is administered at the dose of 3.7 MBq (+/- 10%), once every 8-10 weeks for a planned 4 cycles..

Post-Treatment Follow-up (Safety & Efficacy): Following treatment cessation, all participants will undergo safety follow-up, including a 30-day safety follow-up visit (FUP) and longer-term safety follow-up assessments over approximately 12 months.

Survival Follow-up: After discontinuation of study treatment or completion of the post-treatment follow-up period, participant status will be collected every 90 days (through telephone) as part of survival follow-up. Every effort should be made to adhere to the survival follow-up schedule to ensure collection of survival data. Survival follow-up and the study will conclude when the number of OS events required for the final OS analysis is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic Castration-Resistant Prostate Cancer (mCRPC) mCRPC refers to prostate cancer that progresses despite serum testosterone at castrate levels (< 50 ng/dL or 1.7 nmol/L), meeting at least one of the following criteria:

   * PSA >1 ng/mL with two consecutive rises at least 1 week apart, each increase ≥50% above the nadir.

     * Radiographic progression: Either two or more new bone lesions on bone scan, or soft tissue lesion progression as per RECIST 1.1 criteria. Progression based on symptoms alone is insufficient for mCRPC diagnosis and requires further evaluation.
2. Failure of, Refusal of, Absence of, or Refractoriness to Standard Therapy, or Disease Progression, or No Available Standard Therapy per Current Guidelines:

   * Patients who have not received, refused, or progressed after receiving at least 1 but no more than 2 prior taxane-based therapies. The taxane regimen must have included exposure for at least 2 cycles. Patients who received only one taxane may be included if the investigator deems them unsuitable for a second taxane (e.g., due to frailty assessed by geriatric/comorbidity evaluation or intolerance).

     * Patients who have progressed after receiving at least one novel androgen axis drug [NAAD] (e.g., abiraterone, enzalutamide).
3. Ability to understand and voluntarily sign a written informed consent form (ICF), and willingness and ability to comply with trial procedures including examinations and follow-up.
4. Age 18-90 years (inclusive).
5. Expected survival > 6 months.
6. ECOG performance status ≤ 2.
7. Presence of high-uptake lesions confirmed by 68Ga-PSMA-11 PET/CT imaging (positive defined as lesion uptake >1.5 times the liver background).
8. At least one measurable lesion per RECIST 1.1 criteria OR at least one bone metastasis per PCWG3 criteria.
9. Adequate organ function (No blood products, growth factors, or albumin administered within 14 days prior to baseline lab tests):

   * Bone Marrow Function: Neutrophil count ≥ 1.5 × 10⁹/L, White blood cell count ≥ 3.0 × 10⁹/L, Platelet count ≥ 100 × 10⁹/L, Hemoglobin ≥ 10 g/dL (≥ 100 g/L).

     * Liver Function: Albumin ≥ 30 g/L, Total bilirubin ≤ 1.5 × ULN, ALT or AST ≤ 3.0 × ULN (without liver metastases) or ≤ 5.0 × ULN (with liver metastases).

       * Renal Function: Serum creatinine ≤ 1.5 × ULN.

         * Coagulation: INR ≤ 1.5; Activated partial thromboplastin time (APTT) ≤ 2 × ULN (for patients not on anticoagulation or on stable-dose anticoagulation).
10. Agreement to comply with prescribed radiation protection measures during the trial period.

Exclusion Criteria:

1. Inability to tolerate imaging procedures;
2. Patients who have received systemic anticancer therapy (e.g., chemotherapy, radiotherapy, immunotherapy; excluding endocrine therapy), investigational drugs, or device therapy within 4 weeks prior to dosing;
3. Patients who received radionuclide therapy (Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, Lutetium-177) within 6 months, or any External Beam Radiation Therapy (EBRT) within 2 months prior to the first dose;
4. Patients with unresolved Grade 4 myelosuppression from prior anticancer therapy within 2 weeks, or Grade 3 myelosuppression requiring >6 weeks for recovery;
5. Planned use of cytotoxic chemotherapy, antitumor immunotherapy, radioligand therapy, or similar agents during the study;
6. Use of blood products or albumin within 14 days before dosing to meet enrollment criteria;
7. Brain metastasis at screening, except:

   * Asymptomatic cases confined to supratentorial/cerebellar regions (no midbrain/pons/medulla/spinal cord involvement) without corticosteroid therapy and with lesions ≤1.5 cm;

     * Symptomatic cases with treated and radiologically stable lesions (>4 weeks);
8. Other malignancies within 5 years (excluding cured localized cancers like basal/squamous cell skin carcinoma);
9. Superscan on bone scintigraphy;
10. Symptomatic or impending spinal cord compression;
11. Prior EBRT involving extensive bone marrow (>25%);
12. Significant cardiac disease at screening, including:

    * QTcF >470 ms or long QT syndrome history;

      * Myocardial infarction, angina, or CABG within 6 months deemed ineligible by investigators;
13. Any condition that, per investigator judgment, may compromise safety, data interpretation, or indicate high risk;
14. Uncontrolled bladder outlet obstruction, urinary incontinence, claustrophobia, or radiophobia at screening;
15. Positive for HCV-Ab, HIV, or syphilis antibodies at screening;
16. HBsAg-positive patients with active HBV replication (confirmed by HBV-DNA per investigator assessment);
17. Known allergy to proteins/peptides, excipients, or structurally related compounds;
18. History of drug/alcohol abuse within 1 year or chronic substance abuse;
19. Failure to use effective contraception during the trial and for 6 months post-last dose;
20. Severe active infection prior to the first administration.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen 50 (PSA50) response | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  PSA50 response is defined as the proportion of patients who have a more/equal 50% decrease in PSA from baseline, it will be calculated at 12, 24 and 48 months
Number of participants with Treatment Emergent Adverse Events | From enrollment till 30 days safety follow-up, assessed up to 50 months (estimated final OS analysis)
  The distribution of adverse events (AE) will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of enrollment until date of progression or date of death from any cause, whichever come first, assessed up to 50 months (estimated final OS analysis)
  PSA-PFS is defined as the time from date of enrollment to the date of first documented progression by investigator assessment (radiographic progression, clinical progression, PSA progression) or death from any cause, whichever occurs first
Overall Survival (OS) | From date of enrollment until date of death from any cause, assessed up to 50 months (estimated final OS analysis)
  OS is defined as time to death for any cause

OTHER OUTCOMES:
Time to Response (TTR) | From date of enrollment till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  TTR is defined as the time from the date of enrollment to the date of first documented response (CR or PR).
European Quality of Life ( EuroQoL) -5 Domain 5 Level Scale (EQ-5D-5L) | From screening up till 30 day safety follow-up or week 48 of long term follow up for patient prematurely discontinued, assessed up to 50 months (estimated final OS analysis)
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Study Chair — Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China